#### STUDY PROTOCOL

# **Comparison of Nasal Endotracheal Tube and Spiral Tube for**

### **Nasotracheal Intubation in Pediatric Patients**

06/ May /2025

## **Patient Characteristics**

Patient Name/Surname

Protocol no:

Age/Sex:

Height / Weight / BMI:

**ASA Score:** 

Other diseases:

## **Intubation Data:**

Type of tube and tube number:

NPT / ST No:

**İntubation Time:** 

Number of attempts:

Cormack Lehane Score:

Use of Magill Forceps: Y/N
Video Laryngoscope Usage : Y/N
Sellick Maneuver: Y/N

# **Epistaxis Severity**

## 0. Minute:

- 0 Absent
- 1 Mild
- 2 Moderate
- 3 Severe

### 5. Minute:

- 0 Absent
- 1 Mild
- 2 Moderate
- 3 Severe

# STATISTICAL ANALYSIS

Statistical analyses will be performed using SPSS Statistics for Windows, Version 22.0 software (IBMCorp., Armonk, NY, USA). Statistical analysis will be performed for patient data including descriptive statistics, frequency and other characteristics for all categories. Continuous data will be expressed as mean  $\pm$  standard deviation. Continuous variables will be analyzed with Shapiro-Wilk and Kolmogorov-Smirnov tests to determine whether the data conform to normal distribution. Continuous and normally distributed variables will be compared using Student T-test. Nonparametric tests will be selected when the data are not normally distributed. Categorical variables will be compared using the chi-square test. All p values will be two-sided and p $\leq$ 0.05 will be considered statistically significant.

G power calculation was made by considering similar studies and the power of the study was calculated as 80%.

# **INFORMED CONSENT**

I was informed by Specialist Dr. Zülfü Savaş that a medical research titled "Random Comparison of Nasal Endotracheal Tube and Spiral Tube for Nasotracheal Intubation in Pediatric Patients" would be conducted at Dicle University Faculty of Dentistry and the above information about this research was conveyed to me. After this information, I was invited to participate in such a study as a "participant".

If I participate in this study, I believe that the confidentiality of my personal information, which should remain between me and the physician, will be treated with great care and respect during this research. I have been given sufficient confidence that my personal information will be carefully protected during the use of the research results for educational and scientific purposes. I can withdraw from the study without giving any reason during the conduct of the study (However, I am aware that it would be appropriate to inform the researchers in advance that I will withdraw from the study in order not

to leave them in a difficult situation) Also, provided that no harm is done to my medical condition, the researcher I may be excluded from the research.

I do not assume any financial responsibility for the expenses to be incurred for the research. I will not be paid. I have been given the necessary assurance that any medical intervention will be provided in case of any health problem that may arise, whether directly or indirectly, due to reasons arising from the research application. (I will not be under any financial burden regarding these medical interventions).

If I encounter a health problem during the research, I know that I can reach Specialist Dr. Zülfü Savaş at any time at the phone number 0531 7013696 (mobile) and on the Dicle University Faculty of Dentistry. I do not have to participate in this research and I may not participate. I have not encountered any coercive behavior about my participation in the research. I also know that if I refuse to participate, this will not harm my medical care and my relationship with the physician. I have understood all the explanations given to me in detail. After a period of reflection on my own, I have decided to take part as a "participant" in this research project. I accept the invitation with great pleasure and willingness.

I will receive a copy of this signed form sheet.
Participant
Name, surname:
Address
Tel.
Signature